CLINICAL TRIAL: NCT03863288
Title: Dose-Response Relationship and Pharmacokinetics of Intranasal Oxytocin on Neural Impact in Youth With High Levels of Irritability
Brief Title: Dose Response Relationship of Oxytocin on Irritability in Youths
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per DSMB's recommendation
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0219-20-FB; 1U01MH120155-01A1 (NIH)
Record Dates: First submitted 2018-09-25; First posted 2019-03-05 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Irritable Mood
Keywords: oxytocin; neuroimaging; irritability; fMRI; pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects are randomly assigned to one of 4 doses of OXT or placebo. Investigators and subjects and parents/guardians are blinded to assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Intranasal Spray Placebo (Placebo Comparator): Nasal spray of placebo liquid solution as a single dose. fMRI scan pre and post-administration.
  Interventions: Procedure: Functional MRI (fMRI); Drug: Placebo
- Oxytocin Intranasal Spray 8 International Unit (IU) (Active Comparator): Nasal spray of Oxytocin 8 International Unit (8IU) liquid solution as a single dose. fMRI scan pre and post administration.
  Interventions: Procedure: Functional MRI (fMRI); Drug: Oxytocin Intranasal Spray 8 International Unit (8IU)
- Oxytocin Intranasal Spray 24 International Unit (IU) (Active Comparator): Nasal spray of Oxytocin 24 International Unit (24IU) liquid solution as a single dose. fMRI scan pre and post administration.
  Interventions: Procedure: Functional MRI (fMRI); Drug: Oxytocin intranasal spray 24 International Unit (24IU)
- Oxytocin Intranasal Spray 48 International Unit (IU) (Active Comparator): Nasal spray of Oxytocin 48 International Unit (48IU) liquid solution as a single dose. fMRI scan pre and post administration.
  Interventions: Procedure: Functional MRI (fMRI); Drug: Oxytocin intranasal spray 48 International Unit (48IU)
- Oxytocin Intranasal Spray 80 International Unit (IU) (Active Comparator): Nasal spray of Oxytocin 80 International Unit (80IU) liquid solution as a single dose. fMRI scan pre and post-administration.
  Interventions: Procedure: Functional MRI (fMRI); Drug: Oxytocin intranasal spray 80 International Unit (80IU)

INTERVENTIONS:
Procedure: Functional MRI (fMRI) — Functional MRI (fMRI) scan with affective/cognitive tasks
Drug: Oxytocin Intranasal Spray 8 International Unit (8IU) — Oxytocin intranasal spray liquid administration
  Arms: Oxytocin Intranasal Spray 8 International Unit (IU)
Drug: Oxytocin intranasal spray 24 International Unit (24IU) — Oxytocin intranasal spray liquid administration
  Arms: Oxytocin Intranasal Spray 24 International Unit (IU)
Drug: Oxytocin intranasal spray 48 International Unit (48IU) — Oxytocin intranasal spray liquid administration
  Arms: Oxytocin Intranasal Spray 48 International Unit (IU)
Drug: Oxytocin intranasal spray 80 International Unit (80IU) — Oxytocin intranasal spray liquid administration
  Arms: Oxytocin Intranasal Spray 80 International Unit (IU)
Drug: Placebo — Placebo intranasal spray liquid administration
  Arms: Intranasal Spray Placebo

SUMMARY:
The proposed study is a randomized, double-blind proof of concept (PoC) study on the neural impact of intranasal oxytocin (OXT) administration for adolescents (age 14 to 18), demonstrating a clinically significant level of irritability as defined by a score of ≥4 on the Affective Reactivity Index (ARI). Planned enrollment is 80 subjects over 3 years.

DETAILED DESCRIPTION:
Endogenous oxytocin (OXT) has been a focus of prior psychiatric research due to its role in pro-social behavior, and modulation of response to social/emotional stimuli. Although many studies argue that the intranasal administration of OXT can produce behavioral as well as neural changes, there is surprisingly little comprehensive research on this issue. Most of the previous studies are limited by using a single dose of intranasal OXT in small samples, and there is no current consensus regarding appropriate dosage and very little data on neural impact as a function of dose. There has been little consideration of the relation between pharmacokinetics (peripheral level of OXT after administration) and the degree of induced neural changes. None of these issues have been studied in a pediatric population with clinically significant psychopathology. This study is proposed to determine the extent to which neural changes are induced by OXT intranasal administration, by examining the dose-response relationship (the degree of neural changes induced by various doses of OXT) and the correlation of pharmacokinetics (peripheral level of OXT after administration and the induced neural changes) in youths with clinically significant psychopathology. The form of psychopathology targeted is irritability: the increased propensity to exhibit anger relative to peers.One of the neurobiological mechanisms of irritability implicates dysfunction in the acute threat response system. OXT, with its most commonly proposed mechanism being reduction of hyperactivity in the acute threat response system, is a potentially promising agent to induce neural changes in the target brain areas of the acute threat response system for youths with high levels of irritability. The study aims to quantify the extent to which different doses of OXT will reduce the activation of the acute threat response system to emotional stimuli in youths with high levels of irritability. Both resting state and task-based functional MRI will be used , using affective-cognitive tasks (to obtain the primary aim will begin after the clinician scan) with demonstrated test-retest reliability and capability of capturing the core target areas of OXT administration in the acute threat response system. Pharmacokinetics (plasma and saliva level) after OXT administration will be examined to determine correlation with the induced neural changes in the target areas.

ELIGIBILITY:
Inclusion Criteria:

* 14-18 years of age
* current diagnosis of Attention Deficit/Hyperactivity Disorder (ADHD), Oppositional Defiant Disorder (ODD), Conduct Disorder (CD), or Disruptive Mood Dysregulation Disorder (DMDD) as determined by the Kiddie-Schedule for Affective Disorders and Schizophrenia (K-SADS), lifetime version;54
* Clinically significant level of irritability as defined by a score of ≥4 on the Affective Reactivity Index (ARI)
* If currently on medication, treatment must be stable for at least 2 weeks with stimulant medication, and at least 4 weeks with alpha 2 agonist, atomoxetine, antipsychotics, mood stabilizers, or antidepressant.

Exclusion Criteria:

* Comorbid psychotic, tic, autism spectrum disorder, or substance use disorders, or current diagnosis of bipolar disorder; -Major medical illness that prohibits OXT administration (e.g., severe liver disease, seizure disorder, metabolic disorder)
* Past history of allergic reaction to OXT and its intranasal product
* History of Central Nervous System (CNS) disease (including history of seizure, epilepsy, CNS tumor, CNS hemorrhage, or serious CNS infection including meningitis or encephalitis)
* A positive urine pregnancy test
* A positive urine drug screen or currently active diagnosis of substance use disorder
* Wechsler Abbreviated Scale of Intelligence (WASI-2; two subset form) scores <70
* Metal in the body (i.e., hearing aid, cardiac pacemaker, bone plates, braces, non-removable piercing/implants, etc.), claustrophobia, or any other condition that would preclude MRI scanning.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) response within rostro-medial prefrontal cortex ( rmPFC) region of interest to emotional stimuli during the Affective Stroop (AS) at approximately 50 minutes after intranasal administration of OXT. | 50 minutes
  Neural changes observable on fMRI as BOLD responses in medial prefrontal cortex. Response data will be generated for each participant for the four OXT doses (8, 24, 48 and 80 IU) and placebo.
Plasma concentrations of OXT at 10, 20, 30, 40, and 50 minutes post intranasal OXT administration, and immediately post-fMRI scanning. | 50 minutes and 2 hours
  Area under the curve (OXT dose response)

SECONDARY OUTCOMES:
BOLD responses within the amygdala region of interest (ROI) to emotional stimuli during the Affective Stroop (AS) task (at approximately 50 minutes after intranasal administration of OXT (placebo, 8, 24, 48, and 80 IU). | 50 minutes
  Neural changes observable on fMRI as BOLD responses in amygdala.
The degree of functional connectivity between rmPFC and amygdala during resting-state fMRI (rs-fMRI) after intranasal administration of OXT. | 60 minutes
  functional connectivity observable on rs-fMRI
BOLD responses within peri-aqueductal gray (PAG) and amygdala regions of interest (ROIs) to emotional stimuli during the facial expression task (at approximately 70 minutes) after intranasal administration of OXT. | 70 minutes
  Neural changes observable on fMRI as BOLD responses in PAG and amygdala.
Saliva level of OXT at 10, 20, 30, 40 and 50 minutes post-administration of intranasal OXT, and immediately after fMRI scanning to calculate area under curve (AUC) | 50 minutes and 2 hours
  Area under curve (OXT dose response)

CONTACTS AND LOCATIONS:
Overall Officials: Soonjo Hwang, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Department of Psychiatry, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee MR, Scheidweiler KB, Diao XX, Akhlaghi F, Cummins A, Huestis MA, Leggio L, Averbeck BB. Oxytocin by intranasal and intravenous routes reaches the cerebrospinal fluid in rhesus macaques: determination using a novel oxytocin assay. Mol Psychiatry. 2018 Jan;23(1):115-122. doi: 10.1038/mp.2017.27. Epub 2017 Mar 14. PMID 28289281
- [Background] Beard R , Singh N , Grundschober C , Gee AD , Tate EW . High-yielding 18F radiosynthesis of a novel oxytocin receptor tracer, a probe for nose-to-brain oxytocin uptake in vivo. Chem Commun (Camb). 2018 Jul 17;54(58):8120-8123. doi: 10.1039/c8cc01400k. PMID 29974895
- [Background] Cochran DM, Fallon D, Hill M, Frazier JA. The role of oxytocin in psychiatric disorders: a review of biological and therapeutic research findings. Harv Rev Psychiatry. 2013 Sep-Oct;21(5):219-47. doi: 10.1097/HRP.0b013e3182a75b7d. PMID 24651556
- [Background] Kendrick KM, Guastella AJ, Becker B. Overview of Human Oxytocin Research. Curr Top Behav Neurosci. 2018;35:321-348. doi: 10.1007/7854_2017_19. PMID 28864976
- [Background] Bos PA, Panksepp J, Bluthe RM, van Honk J. Acute effects of steroid hormones and neuropeptides on human social-emotional behavior: a review of single administration studies. Front Neuroendocrinol. 2012 Jan;33(1):17-35. doi: 10.1016/j.yfrne.2011.01.002. Epub 2011 Jan 21. PMID 21256859
- [Background] Insel TR. Translating Oxytocin Neuroscience to the Clinic: A National Institute of Mental Health Perspective. Biol Psychiatry. 2016 Feb 1;79(3):153-4. doi: 10.1016/j.biopsych.2015.02.002. Epub 2015 Nov 16. No abstract available. PMID 26723108
- [Background] Spengler FB, Schultz J, Scheele D, Essel M, Maier W, Heinrichs M, Hurlemann R. Kinetics and Dose Dependency of Intranasal Oxytocin Effects on Amygdala Reactivity. Biol Psychiatry. 2017 Dec 15;82(12):885-894. doi: 10.1016/j.biopsych.2017.04.015. Epub 2017 May 10. PMID 28629540
- [Background] Striepens N, Kendrick KM, Hanking V, Landgraf R, Wullner U, Maier W, Hurlemann R. Elevated cerebrospinal fluid and blood concentrations of oxytocin following its intranasal administration in humans. Sci Rep. 2013 Dec 6;3:3440. doi: 10.1038/srep03440. PMID 24310737
- [Background] Netherton E, Schatte D. Potential for oxytocin use in children and adolescents with mental illness. Hum Psychopharmacol. 2011 Jun-Jul;26(4-5):271-81. doi: 10.1002/hup.1212. Epub 2011 Jul 12. PMID 21751251
- [Background] Leibenluft E. Pediatric Irritability: A Systems Neuroscience Approach. Trends Cogn Sci. 2017 Apr;21(4):277-289. doi: 10.1016/j.tics.2017.02.002. Epub 2017 Mar 6. PMID 28274677
- [Background] Blair RJR. Traits of empathy and anger: implications for psychopathy and other disorders associated with aggression. Philos Trans R Soc Lond B Biol Sci. 2018 Apr 19;373(1744):20170155. doi: 10.1098/rstb.2017.0155. PMID 29483341
- [Background] Grace SA, Rossell SL, Heinrichs M, Kordsachia C, Labuschagne I. Oxytocin and brain activity in humans: A systematic review and coordinate-based meta-analysis of functional MRI studies. Psychoneuroendocrinology. 2018 Oct;96:6-24. doi: 10.1016/j.psyneuen.2018.05.031. Epub 2018 May 24. PMID 29879563
- [Background] Leibenluft E, Stoddard J. The developmental psychopathology of irritability. Dev Psychopathol. 2013 Nov;25(4 Pt 2):1473-87. doi: 10.1017/S0954579413000722. PMID 24342851
- [Background] Wiggins JL, Brotman MA, Adleman NE, Kim P, Oakes AH, Reynolds RC, Chen G, Pine DS, Leibenluft E. Neural Correlates of Irritability in Disruptive Mood Dysregulation and Bipolar Disorders. Am J Psychiatry. 2016 Jul 1;173(7):722-30. doi: 10.1176/appi.ajp.2015.15060833. Epub 2016 Feb 19. PMID 26892942
- [Background] Hwang S, Nolan ZT, White SF, Williams WC, Sinclair S, Blair RJ. Dual neurocircuitry dysfunctions in disruptive behavior disorders: emotional responding and response inhibition. Psychol Med. 2016 May;46(7):1485-96. doi: 10.1017/S0033291716000118. Epub 2016 Feb 15. PMID 26875722
- [Background] Hwang S, White SF, Nolan ZT, Sinclair S, Blair RJ. Neurodevelopmental changes in the responsiveness of systems involved in top down attention and emotional responding. Neuropsychologia. 2014 Sep;62:277-85. doi: 10.1016/j.neuropsychologia.2014.08.003. Epub 2014 Aug 13. PMID 25128588
- [Background] Leppanen J, Ng KW, Kim YR, Tchanturia K, Treasure J. Meta-analytic review of the effects of a single dose of intranasal oxytocin on threat processing in humans. J Affect Disord. 2018 Jan 1;225:167-179. doi: 10.1016/j.jad.2017.08.041. Epub 2017 Aug 17. PMID 28837950
- [Background] Koch SB, van Zuiden M, Nawijn L, Frijling JL, Veltman DJ, Olff M. Intranasal Oxytocin Administration Dampens Amygdala Reactivity towards Emotional Faces in Male and Female PTSD Patients. Neuropsychopharmacology. 2016 May;41(6):1495-504. doi: 10.1038/npp.2015.299. Epub 2015 Sep 25. PMID 26404844
- [Background] Wakschlag LS, Estabrook R, Petitclerc A, Henry D, Burns JL, Perlman SB, Voss JL, Pine DS, Leibenluft E, Briggs-Gowan ML. Clinical Implications of a Dimensional Approach: The Normal:Abnormal Spectrum of Early Irritability. J Am Acad Child Adolesc Psychiatry. 2015 Aug;54(8):626-34. doi: 10.1016/j.jaac.2015.05.016. Epub 2015 Jun 14. PMID 26210331
- [Background] Eckstein M, Markett S, Kendrick KM, Ditzen B, Liu F, Hurlemann R, Becker B. Oxytocin differentially alters resting state functional connectivity between amygdala subregions and emotional control networks: Inverse correlation with depressive traits. Neuroimage. 2017 Apr 1;149:458-467. doi: 10.1016/j.neuroimage.2017.01.078. Epub 2017 Feb 1. PMID 28161309
- [Background] Wynn JK, Green MF, Hellemann G, Reavis EA, Marder SR. A dose-finding study of oxytocin using neurophysiological measures of social processing. Neuropsychopharmacology. 2019 Jan;44(2):289-294. doi: 10.1038/s41386-018-0165-y. Epub 2018 Jul 28. PMID 30082892
- [Background] Lefevre A, Mottolese R, Dirheimer M, Mottolese C, Duhamel JR, Sirigu A. A comparison of methods to measure central and peripheral oxytocin concentrations in human and non-human primates. Sci Rep. 2017 Dec 8;7(1):17222. doi: 10.1038/s41598-017-17674-7. PMID 29222505
- [Background] Hwang S, White SF, Nolan ZT, Craig Williams W, Sinclair S, Blair RJ. Executive attention control and emotional responding in attention-deficit/hyperactivity disorder--A functional MRI study. Neuroimage Clin. 2015 Oct 9;9:545-54. doi: 10.1016/j.nicl.2015.10.005. eCollection 2015. PMID 26640766
- [Background] White SF, Marsh AA, Fowler KA, Schechter JC, Adalio C, Pope K, Sinclair S, Pine DS, Blair RJ. Reduced amygdala response in youths with disruptive behavior disorders and psychopathic traits: decreased emotional response versus increased top-down attention to nonemotional features. Am J Psychiatry. 2012 Jul;169(7):750-8. doi: 10.1176/appi.ajp.2012.11081270. PMID 22456823